CLINICAL TRIAL: NCT03111043
Title: Head-to-pelvis Computed Tomography Evaluation of Sudden Death Survivors
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Medic One Foundation (Other); Harborview Injury Prevention and Research Center (Other)
Responsible Party: Principal Investigator, Kelley Branch, Professor, Medicine/Cardiology, University of Washington
Other Study IDs: STUDY00001380
Record Dates: First submitted 2017-03-24; First posted 2017-04-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Sudden Death; Out-Of-Hospital Cardiac Arrest
Keywords: computed tomography; Sudden cardiac arrest; Cardiac computed tomography; Diagnostic accuracy; Clinical outcome
MeSH Terms: conditions — Death, Sudden; Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Head to pelvis CT scan — Introduction of early head to pelvis CT scan within 6 hours of out of hospital arrest as an adjunct to standard of care (no randomization)

SUMMARY:
Out-of-hospital arrest can occur from multiple etiologies. In patients without an obvious reason for the sudden-death event, diagnostic evaluation is not clear. This study is to determine if early imaging with a head-to-pelvis CT scan may improve diagnostic accuracy, speed of diagnosis and potentially clinical outcomes.

DETAILED DESCRIPTION:
Best practices for survivors of out-of-hospital sudden death are underdeveloped and untested. Early diagnosis in sudden death survivors is challenging due to patient intubation and obtundation, limited history, and imprecise standard of care testing. Sudden death without an obvious cause (termed "idiopathic sudden death") is primarily caused by cardiovascular disease although a large number of cases result from non-cardiac disease. Improvements in computed tomography (CT) technologies provides a means to identify up to 86% of idiopathic causes of sudden death, including cardiovascular and coronary artery disease, cerebral disease, pulmonary embolism and abdominal catastrophe4 as well as secondary injury from cardiopulmonary resuscitation. To date, use of early CT scans on consecutive sudden death survivors has not been reported. The innovation of this pilot trial is to be first to test whether a comprehensive head-to-pelvis, ECG-gated contrast CT scan (CT-First) can identify the majority of causes for idiopathic sudden death. The significance of CT-First approach is potentially reducing diagnostic errors, treatment delays and inappropriate treatments to potentially improve clinical outcomes in this very high risk population. The expertise of the medical centers involved, combined with the highly respected Medic One service, provide an unusual opportunity to test this diagnostic paradigm with cutting edge CT technologies. The data generated from this study will be used to plan larger randomized trials of early contrast CT scanning versus invasive coronary angiography in sudden death survivors and may be extrapolated to other patient populations such as possible acute coronary syndrome or after trauma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients reaching the Emergency Department within 6 hours of resuscitated sudden death.
2. No obvious cause for sudden death event with initial standard of care clinical evaluation
3. Clinically stable to have CT performed per treating physician
4. Candidates for continued intubation and sedation during the CT scan with or without therapeutic hypothermia protocol.

Exclusion Criteria:

1. Meets criteria for acute ST elevation myocardial infarction (ST elevation ≥1 contiguous lead or new or unknown duration left bundle branch block on ECG) or has other indication for ICA
2. Obvious cause of sudden death - Examples: witnessed trauma, drowning, suicide attempt
3. Known non-revascularized coronary artery disease or coronary stent <2.5 mm.
4. Known severe renal dysfunction (eGFR<30 ml/hr, creatinine >1.7 mg/dl)
5. Implantable defibrillator, due to metal artifact from defibrillator coil
6. Known iodinated contrast allergy
7. Known hospice patient or terminal disease with expected <3 months survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals in the Seattle Fire Department or King County, Washington Emergency Medical Services service area
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy compared to adjudicated diagnosis for sudden-death event | During hospitalization (up to 6 months)
Time to correct diagnosis by head to pelvis CT scan | During hospitalization (up to 6 months)
Cost analysis of head to pelvis CT scan - payer perspective | During hospitalization (up to 6 months)

SECONDARY OUTCOMES:
Determine adjudicated causes for sudden-death event in survivors | During hospitalization (up to 6 months)
Clinical outcomes for sudden-death survivors undergoing head to pelvis CT scan | During hospitalization (up to 6 months)
  Clinical outcomes include in-hospital survival, circulatory arrest, survival to discharge, and discharge status (discharge to home, nursing facility)
Determine complications of cardiopulmonary resuscitation on thoracoabdominal organs measured by CT in sudden death survivors | During hospitalization (up to 6 months)

OTHER OUTCOMES:
Safety outcome: Incidence of contrast associated acute kidney injury. | 48 hours from CT scan (up to 6 months)
Safety outcome: Prevalence of false positive CT findings leading to incorrect treatment | During hospitalization (up to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Branch, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Unclear plan for sharing data.

REFERENCES:
- [Background] Branch KRH, Strote J, Gunn M, Maynard C, Kudenchuk PJ, Brusen R, Petek BJ, Sayre MR, Edwards R, Carlbom D, Counts CR, Probstfield JL, Gatewood MO. Early head-to-pelvis computed tomography in out-of-hospital circulatory arrest without obvious etiology. Acad Emerg Med. 2021 Apr;28(4):394-403. doi: 10.1111/acem.14228. Epub 2021 Mar 24. PMID 33606342
- [Background] Branch KR, Hira R, Brusen R, Maynard C, Kudenchuk PJ, Petek BJ, Strote J, Sayre MR, Gatewood M, Carlbom D, Counts C, Probstfield JL, Gunn M. Diagnostic accuracy of early computed tomographic coronary angiography to detect coronary artery disease after out-of-hospital circulatory arrest. Resuscitation. 2020 Aug;153:243-250. doi: 10.1016/j.resuscitation.2020.04.033. Epub 2020 May 15. PMID 32422241
- [Background] Karatasakis A, Sarikaya B, Liu L, Gunn ML, Kudenchuk PJ, Gatewood MO, Maynard C, Sayre MR, Counts CR, Carlbom DJ, Edwards RM, Branch KRH. Prevalence and Patterns of Resuscitation-Associated Injury Detected by Head-to-Pelvis Computed Tomography After Successful Out-of-Hospital Cardiac Arrest Resuscitation. J Am Heart Assoc. 2022 Feb;11(3):e023949. doi: 10.1161/JAHA.121.023949. Epub 2022 Jan 19. PMID 35043689
- [Background] Branch KRH, Gatewood MO, Kudenchuk PJ, Maynard C, Sayre MR, Carlbom DJ, Edwards RM, Counts CR, Probstfield JL, Brusen R, Johnson N, Gunn ML. Diagnostic yield, safety, and outcomes of Head-to-pelvis sudden death CT imaging in post arrest care: The CT FIRST cohort study. Resuscitation. 2023 Jul;188:109785. doi: 10.1016/j.resuscitation.2023.109785. Epub 2023 Apr 3. PMID 37019352